CLINICAL TRIAL: NCT01880424
Title: A Phase 3, International, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group Efficacy and Safety Trial of Linaclotide Administered Orally for 12 Weeks to Patients With Irritable Bowel Syndrome With Constipation (IBS-C)
Acronym: D5630C00001
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Ironwood Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ICP-103-307
Record Dates: First submitted 2013-06-12; First posted 2013-06-19 (Estimated); Results first posted 2016-09-27 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-08

CONDITIONS: Irritable Bowel Syndrome With Constipation (IBS-C)
MeSH Terms: interventions — linaclotide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- controlled arm (Placebo Comparator)
  Interventions: Drug: Placebo
- treatment arm (Experimental)
  Interventions: Drug: Linaclotide

INTERVENTIONS:
Drug: Placebo — matching Placebo Capsules, Oral, once daily
  Arms: controlled arm
Drug: Linaclotide — Linaclotide 290 ug Capsules, Oral, once daily
  Arms: treatment arm

SUMMARY:
This clinical trial is an international, multicenter, randomized, double-blind, placebo-controlled, parallel-group trial comparing one dose of linaclotide to placebo. Approximately 800 patients with a diagnosis of IBS-C (modified Rome III criteria) will be randomized at up to 60 trial centers in China, Australia, and New Zealand.

The trial will consist of up to 21 days of screening, 14 to 21 days of pre-treatment, 12 weeks of double-blind treatment, and 2 weeks of follow-up. At the end of the Pre-treatment Period, patients meeting the entry criteria for this trial will be randomized to one of two double-blind treatment groups: 290 ug linaclotide, or placebo (1:1).

ELIGIBILITY:
Inclusion Criteria:

1. Patient has signed an Informed Consent Form(ICF).
2. Patient Must not be pregnant or breastfeeding and agree to use birth control
3. Patient meets the colonoscopy requirements defined by the American Gastroenterological Association guidelines and no clinically-significant laboratory or physical examination findings;
4. Patient meets protocol-defined criteria for Irritable Bowel Syndrome with Constipation(IBS-C), including stool frequency, straining, stool consistency, abdominal pain, and abdominal discomfort criteria
5. Patient meets protocol-defined eDiary completion Compliance and agrees to refrain from making any new, major life-style changes that may affect IBS-C symptoms

Exclusion Criteria:

1. Recent history of mushy or watery stools
2. Various medical conditions, medical histories, or family medical histories that would not make the patient a good candidate for the study
3. Patient currently has both unexplained and clinically significant alarm symptoms or systemic signs of infection or colitis.
4. Surgery to the gastrointestinal tract
5. Usage of prohibited medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1722 (Actual)
Dates: Start 2013-07; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yunsheng Yang, Principal Investigator — Chinese PLA General Hospital; Shutian Zhang, Principal Investigator — Beijing Friendship Hospital; Zhaoshen Li, Principal Investigator — Changhai Hospital Affiliated to Second Military Mecical University of Chinese PLA; Weifen Xie, Principal Investigator — Changzheng Hospital Affiliated to Second Military Mecical University of Chinese PLA; Yaozong Yuan, Principal Investigator — Ruijin Hospital Affiliated to Medical College of Shanghai Jiaotong University; Youqing Xu, Principal Investigator — Beijing Tiantan Hospital; Dongfeng Chen, Principal Investigator — The Third Affiliated Hospital of Third Military Mecical University of Chinese PLA; Minhu Chen, Principal Investigator — The First Affiliated Hospital, Zhongshan (Sun Yat-sen) University; Yanqing Li, Principal Investigator — Qilu Hospital of Shandong University; Xiaozhong Guo, Principal Investigator — General Hospital of Shenyang Military Region of Chinese PLA; Youlin Yang, Principal Investigator — First Affiliated Hospital of Harbin Medical University; Rongquan Wang, Principal Investigator — The First Affiliated Hospital of Third Military Mecical University of Chinese PLA; Xiaohua Hou, Principal Investigator — Union Hospital of Tongji Medical College of Huazhong University of Science & Technology; Liangping Li, Principal Investigator — Sichuang Provincial People's Hospital; Chengwei Tang, Principal Investigator — West China Hospital; Jianlin Ren, Principal Investigator — Zhongshan Hospital Affiliated to Xiamen University; Xizhong Shen, Principal Investigator — Shanghai Zhongshan Hospital; Yulan Liu, Principal Investigator — Peking University People's Hospital; Dongmei Qian, Principal Investigator — Beijing Tongren Hospital Affiliated to Capital Medical University; Huahong Wang, Principal Investigator — Peking University First Hospital
Locations (82):
- United States (52):
  - Research Site, Huntsville, Alabama
  - Research Site, North Little Rock, Arkansas
  - Research Site, Phoenix, Arkansas
  - Research Site, Artesia, California
  - Research Site, Chula Vista, California
  - Research Site, Encino, California
  - Research Site, North Hollywood, California
  - Research Site, Orange, California
  - Research Site, Riverside, California
  - Research Site, San Diego, California
  - Research Site, Boynton Beach, Florida
  - Research Site, Brandon, Florida
  - Research Site, Brooksville, Florida
  - Research Site, Doral, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Kissimmee, Florida
  - Research Site, Lauderdale Lakes, Florida
  - Research Site, Miami, Florida
  - Research Site, Miami Lakes, Florida
  - Research Site, Addison, Illinois
  - Research Site, Evansville, Indiana
  - Research Site, Crowley, Louisiana
  - Research Site, Monroe, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Boston, Massachusetts
  - Research Site, Chesterfield, Michigan
  - Research Site, Wyoming, Michigan
  - Research Site, St Louis, Missouri
  - Research Site, Billings, Montana
  - Research Site, Las Vegas, Nevada
  - Research Site, Brooklyn, New York
  - Research Site, Great Neck, New York
  - Research Site, New York, New York
  - Research Site, Raleigh, North Carolina
  - Research Site, Salisbury, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Franklin, Ohio
  - Research Site, Mentor, Ohio
  - Research Site, Greer, South Carolina
  - Research Site, Chattanooga, Tennessee
  - Research Site, Kingsport, Tennessee
  - Research Site, Knoxville, Tennessee
  - Research Site, Smyrna, Tennessee
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Webster, Texas
  - Research Site, Ogden, Utah
  - Research Site, Lynchburg, Virginia
  - Research Site, Morgantown, West Virginia
- Australia (7):
  - Research Site, Adelaide
  - Research Site, Brisbane
  - Research Site, Five Dock
  - Research Site, Malvern
  - Research Site, Maroubra
  - Research Site, Melbourne
  - Research Site, Parkville
- Research Site, Vaughan, Ontario, Canada
- China (17):
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Harerbin
  - Research Site, Hefei
  - Research Site, Jinan
  - Research Site, Nanchang
  - Research Site, Qingdao
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Shijiazhuang
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Xiamen
- New Zealand (5):
  - Research Site, Auckland
  - Research Site, Christchurch
  - Research Site, Dunedin
  - Research Site, Tauranga
  - Research Site, Wellington

REFERENCES:
- [Derived] Peng LH, Fang JY, Dai N, Shen XZ, Yang YL, Sun J, Yang YS. Efficacy and safety of linaclotide in patients with irritable bowel syndrome with constipation: Chinese sub-cohort analysis of a phase III, randomized, double-blind, placebo-controlled trial. J Dig Dis. 2022 Feb;23(2):99-110. doi: 10.1111/1751-2980.13081. PMID 35019221

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient recruitment occurred over an 18-month period from July 2013 to January 2015 at 98 study centers (40 in China, 42 in the US, 10 in Australia, 5 in New Zealand, and 1 in Canada).
Pre-assignment Details: Patients went through a 14 to 21-day Pretreatment Period during which they provided qualifying bowel habit and symptom severity assessments and rescue medicine usage through an electronic diary (eDiary). 1722 patients provided consents with 839 qualified to join th study.
Groups:
- Linaclotide Arm: Linaclotide 290 ug capsules, oral, once daily
- Placebo Arm: matching placebo capsules, oral, once daily
Period: Overall Study
Arm/Group | Linaclotide Arm | Placebo Arm
Started | 417 | 422
Completed | 384 | 367
Not Completed | 33 | 55
Not completed — Adverse Event | 7 | 6
Not completed — Lack of Efficacy | 1 | 4
Not completed — Lost to Follow-up | 3 | 2
Not completed — Protocol Violation | 11 | 13
Not completed — Withdrawal by Subject | 10 | 30
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent to Treat (ITT) Population (all 839 randomized patients)
Groups:
- Total: Total of all reporting groups
Arm/Group | Linaclotide Arm | Placebo Arm | Total
Number analyzed (Participants) | 417 | 422 | 839
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.0 (13.1) | 41.3 (13.5) | 41.1 (13.3)
Age, Customized [Number; unit: participants]
  between 18 to 65 years | 400 | 405 | 805
  >= 65 years | 17 | 17 | 34
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 333 | 355 | 688
  Male | 84 | 67 | 151
countries [Number; unit: Participants]
  China | 327 | 332 | 659
  Canada | 3 | 3 | 6
  Australia | 19 | 14 | 33
  New Zealand | 4 | 4 | 8
  United States | 64 | 69 | 133

OUTCOME MEASURES:

1. Primary Outcome: 12-week Abdominal Pain/Abdominal Discomfort Weekly Responder
Description: A 12-week Abdominal Pain/Abdominal Discomfort Responder is a patient who meets the Abdominal Pain/Abdominal Discomfort Weekly Responder criteria (i.e., an improvement of ≥30% from baseline in either the mean abdominal pain score or mean abdominal discomfort score for that week, with neither score worsening from baseline for that week) for at least 6 out of the 12 weeks of the Treatment Period.
  Abdominal pain at its worst (in the last 24 hours) was assessed daily by patients on an 11-point numerical rating scale (NRS) where 0 represents no abdominal pain and 10 represents very severe abdominal pain.
  Abdominal discomfort (in the last 24 hours) was assessed daily by patients on an 11-point NRS where 0 represents no abdominal discomfort and 10 represents very severe abdominal discomfort.
Time Frame: Baseline and Weeks 1-12 during the Treatment Period
Population: Intent to Treat (ITT) Population (all 839 randomized patients). If a patient did not have an abdominal pain score or abdominal discomfort score for a particular Treatment Period week, the patient was not considered a responder for that week.
Measure: Number; unit: Participants
Arm/Group | Linaclotide Arm | Placebo Arm
Number analyzed (Participants) | 417 | 422
Participants | 250 | 206
Statistical Analysis 1: Comparison: Linaclotide Arm vs Placebo Arm; Null Hypothesis: There is no difference between the linaclotide dose and placebo in the proportion of 12-week Abdominal Pain/Abdominal Discomfort Responders or there is no difference in the proportion of 12-week IBS Degree of Relief Responders. With 800 planned patients, the statistical power was expected to be approximately 95%, with an overall type I error rate controlled at the 0.05 level (2-sided), based on assumptions from NCT00948818 (LIN-MD-31) study data; Test type: Superiority or Other; p = 0.0010, Cochran-Mantel-Haenszel — Statistical significance (p<0.05) was required in both co-primary efficacy parameters to meet the primary efficacy objective; both p-values met this criterion; Cochran-Mantel-Haenszel test controlling for geographic region; Odds Ratio (OR) = 1.59, 95% CI [1.21 to 2.09] — Odds ratio for response rate (linaclotide : placebo)

2. Primary Outcome: 12-week Irritable Bowel Syndrome (IBS) Degree of Relief Responder
Description: A 12-week IBS Degree of Relief Responder is a patient who meets the IBS Degree of Relief Weekly Responder criteria (i.e., response to the degree of relief of IBS symptoms question for that week was "Considerably relieved" or "Completely relieved") for at least 6 out of the 12 weeks of the Treatment Period.
  Degree of relief of IBS symptoms (in the last 7 days) was assessed weekly by patients on a 7-point balanced ordinal scale where 1 = Completely relieved, 4 = Unchanged, and 7 = As bad as I can imagine.
Time Frame: Baseline and Weeks 1-12 during the Treatment Period
Population: Intent to Treat (ITT) Population (all 839 randomized patients). If a patient did not have an IBS degree of relief score for a particular Treatment Period week, the patient was not considered a responder for that week.
Measure: Number; unit: Participants
Arm/Group | Linaclotide Arm | Placebo Arm
Number analyzed (Participants) | 417 | 422
Participants | 132 | 65
Statistical Analysis 1: Comparison: Linaclotide Arm vs Placebo Arm; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Cochran-Mantel-Haenszel test controlling for geographic region; Odds Ratio (OR) = 2.56, 95% CI [1.83 to 3.58] — Odds ratio for response rate (linaclotide : placebo)

3. Secondary Outcome: Change From Baseline in 12-week Complete Spontaneous Bowel Movement Frequency Rate
Description: The change from baseline in 12-week CSBM frequency (i.e., average weekly CSBM frequency over the 12 weeks of the Treatment Period).
  A spontaneous bowel movement (SBM) is defined as a bowel movement without laxative use in the preceding 24 hours. A CSBM is defined as an SBM that is associated with a sense of complete evacuation.
Time Frame: Baseline and 12-week Treatment Period
Population: Intent to Treat (ITT) Population (all 839 randomized patients); analysis includes patients with analysis values at both baseline and during the Treatment Period. An observed cases approach to missing post-baseline data was applied (i.e., no imputation for missing values).
Measure: Least Squares Mean (Standard Error); unit: CSBMs per Week
Arm/Group | Linaclotide Arm | Placebo Arm
Number analyzed (Participants) | 417 | 422
CSBMs per Week | 1.94 (0.15) | 0.97 (0.15)

4. Secondary Outcome: Change From Baseline in 12-week Spontaneous Bowel Movement Frequency Rate
Description: The change from baseline in 12-week SBM frequency (i.e., average weekly SBM frequency over the 12 weeks of the Treatment Period).
  SBM is defined as a bowel movement without laxative use in the preceding 24 hours.
Time Frame: Baseline and 12-week Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: SBMs per Week
Arm/Group | Linaclotide Arm | Placebo Arm
Number analyzed (Participants) | 417 | 422
SBMs per Week | 2.96 (0.17) | 1.51 (0.17)

5. Secondary Outcome: Change From Baseline in 12-week Stool Consistency
Description: The change from baseline in 12-week stool consistency (i.e., the average of the non-missing Bristol Stool Form Scale [BSFS] score from the SBMs occurring during the 12-week Treatment Period).
  Consistency of each bowel movement was assessed daily by patients using the 7-point BSFS (1=Separate hard lumps like nuts [difficult to pass] to 7=Watery, no solid pieces [entirely liquid]).
Time Frame: Baseline and 12-week Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale (BSFS)
Arm/Group | Linaclotide Arm | Placebo Arm
Number analyzed (Participants) | 371 | 360
Units on a Scale (BSFS) | 1.51 (0.07) | 0.82 (0.07)

6. Secondary Outcome: Change From Baseline in 12-week Severity of Straining
Description: The change from baseline in 12-week severity of straining (i.e., the average of the non-missing straining scores from the SBMs occurring during the 12-week Treatment Period).
  Severity of straining was assessed daily by patients on a 5-point ordinal scale (1=Not at all to 5=An extreme amount).
Time Frame: Baseline and 12-week Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Linaclotide Arm | Placebo Arm
Number analyzed (Participants) | 371 | 360
Units on a Scale | -1.02 (0.05) | -0.69 (0.05)

7. Secondary Outcome: Change From Baseline in 12-week Abdominal Bloating
Description: The change from baseline in 12-week abdominal bloating (i.e., the average of the non-missing daily abdominal bloating scores reported during the 12-week Treatment Period).
  Abdominal bloating (in the last 24 hours) was assessed daily by patients on an 11-point NRS where 0 represents no abdominal bloating and 10 represents very severe abdominal bloating.
Time Frame: Baseline and 12-week Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Linaclotide Arm | Placebo Arm
Number analyzed (Participants) | 417 | 419
Units on a Scale | -1.50 (0.12) | -0.94 (0.12)

8. Secondary Outcome: Change From Baseline in 12-week Abdominal Pain
Description: The change from baseline in 12-week abdominal pain (i.e., the average of the non-missing daily abdominal pain scores reported during the 12-week Treatment Period).
  Abdominal pain at its worst (in the last 24 hours) was assessed daily by patients on an 11-point NRS where 0 represents no abdominal pain and 10 represents very severe abdominal pain.
Time Frame: Baseline and 12-week Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Linaclotide Arm | Placebo Arm
Number analyzed (Participants) | 417 | 419
Units on a Scale | -1.56 (0.12) | -1.07 (0.12)

9. Secondary Outcome: Change From Baseline in 12-week Abdominal Discomfort
Description: The change from baseline in 12-week abdominal discomfort (i.e., the average of the non-missing daily abdominal discomfort scores reported during the 12-week Treatment Period).
  Abdominal discomfort (in the last 24 hours) was assessed daily by patients on an 11-point NRS where 0 represents no abdominal discomfort and 10 represents very severe abdominal discomfort.
Time Frame: Baseline and 12-week Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Linaclotide Arm | Placebo Arm
Number analyzed (Participants) | 417 | 419
Units on a Scale | -1.46 (0.12) | -0.98 (0.12)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from July 2013 to May 2015 (12 weeks of safety data were collected). Includes serious adverse events that occurred on or after the date of the first dose of study drug and within 30 days of the last dose of study drug.
Description: Of the 839 randomized patients, a total of 835 patients received at least one dose of double-blind study drug and were included in the Safety Population.
Arm/Group | Linaclotide Arm | Placebo Arm
Serious Adverse Events (participants affected / at risk) | 4/416 | 10/419
Other Adverse Events (participants affected / at risk) | 56/416 | 26/419
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Linaclotide Arm (N=416) | Placebo Arm (N=419)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Pericoronitis (Infections and infestations) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Multiple system atrophy (Nervous system disorders) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Bladder outlet obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Abortion induced (Surgical and medical procedures) | 1 (1) | 4 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.03% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Linaclotide Arm (N=416) | Placebo Arm (N=419)
Diarrhea (Gastrointestinal disorders) | 39 (39) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 18 (18) | 21 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data generated in this trial will be the property of AstraZeneca and Ironwood Pharmaceuticals, Inc. An integrated clinical and statistical report will be prepared at the completion of the trial. Publication of the results by the Investigator will be subject to mutual agreement between the Investigator, AstraZeneca, and Ironwood Pharmaceuticals, Inc.